CLINICAL TRIAL: NCT02721615
Title: Evaluation of the Potential Adverse Effect of Pressure After Spinal Cord Injury
Brief Title: Injured Spinal Cord Pressure Evaluation
Acronym: ISCoPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: Foundation Wings For Life (Other); Neurosciences Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09.0151; 10/H0807/23 (Registry Identifier: Research ethics commitee - Camberwell St Giles)
Record Dates: First submitted 2016-03-17; First posted 2016-03-29 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Spinal Cord Injuries
Keywords: intra spinal pressure; spinal cord perfusion pressure; microdialysis; duroplasty
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Laminectomy (Active Comparator): Comparison of bone decompression versus no decompression for reducing intra spinal pressure
  Interventions: Procedure: Insertion of intra spinal sub dural pressure monitor
- Duraplasty (Active Comparator): Expansion duraplasty versus no duraplasty for reducing intraspinal pressure
  Interventions: Procedure: Insertion of intra spinal sub dural pressure monitor; Procedure: Insertion of sub dural microdialysis probe
- Hypothermia (Active Comparator): Localised hypothermia for reducing intra spinal pressure and improving spinal cord metabolism
  Interventions: Procedure: Insertion of intra spinal sub dural pressure monitor; Procedure: Insertion of sub dural microdialysis probe

INTERVENTIONS:
Procedure: Insertion of intra spinal sub dural pressure monitor
  Other Names: codman microsensor transducer. Ref. 626638
Procedure: Insertion of sub dural microdialysis probe
  Other Names: CMA61, CMA microdialysis AB. Ref.8010226
  Arms: Duraplasty; Hypothermia

SUMMARY:
About a thousand people a year in the United Kingdom survive a spinal cord injury but are left paralysed or wheelchair-bound. The annual cost of care for spinal cord injury victims is more than half a billion pounds. We propose that after spinal cord injury, cord pressure at the injury site rises, damaging the spinal cord further by secondary ischaemia. The value of measuring and reducing cord pressure after spinal cord injury is unknown.

The injured spinal cord is compressed by bone malalignment and cord swelling. Current management involves realigning and fixing the bony fragments using metal screws, rods and plates. We hypothesise that: 1. Bony realignment alone does not adequately decompress the swollen cord, which remains compressed against the surrounding dura. 2. That duraplasty reduces intra spinal pressure more effectively than bone realignment alone. 3. Localised hypothermia reduces intra spinal pressure and improves metabolism.

We will develop a novel method to measure cord pressure and metabolism at the injury site after spinal cord injury and determine whether the cord pressure rises, for how long, and with what impact on spinal cord metabolism.

This is a pilot study to find out whether spinal cord pressure and metabolism can be measured after spinal cord injury and whether they are effected by treatment choices. We will examine if spinal cord perfusion pressure correlates with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of traumatic spinal cord injury American Spinal Injuries Association grade A-C spinal cord injury Presents within 72hrs of injury Capacity to consent for study

Exclusion Criteria:

Concurrent major co-morbidity likely to influence outcome Other major concurrent injury likely to influence outcome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2024-09 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Intra spinal pressure | 0-7 days
  Intra spinal pressure measured for up to 7 days using sub dural probe
Spinal metabolites | 0-7 days
  Spinal cord metabolites measured using microdialysis probe

CONTACTS AND LOCATIONS:
Overall Officials: Marios C Papadopoulos, MD, Principal Investigator — St George's, University of London
Locations (1):
- St George's, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Werndle MC, Zoumprouli A, Sedgwick P, Papadopoulos MC. Variability in the treatment of acute spinal cord injury in the United Kingdom: results of a national survey. J Neurotrauma. 2012 Mar 20;29(5):880-8. doi: 10.1089/neu.2011.2038. Epub 2011 Oct 26. PMID 21939394
- [Result] Phang I, Mada M, Kolias AG, Newcombe VF, Trivedi RA, Carpenter A, Hawkes RC, Papadopoulos MC. Magnetic Resonance Imaging of the Codman Microsensor Transducer Used for Intraspinal Pressure Monitoring: Findings From the Injured Spinal Cord Pressure Evaluation Study. Spine (Phila Pa 1976). 2016 May;41(10):E605-10. doi: 10.1097/BRS.0000000000001334. PMID 26641852
- [Result] Varsos GV, Werndle MC, Czosnyka ZH, Smielewski P, Kolias AG, Phang I, Saadoun S, Bell BA, Zoumprouli A, Papadopoulos MC, Czosnyka M. Intraspinal pressure and spinal cord perfusion pressure after spinal cord injury: an observational study. J Neurosurg Spine. 2015 Dec;23(6):763-71. doi: 10.3171/2015.3.SPINE14870. Epub 2015 Aug 14. PMID 26273764
- [Result] Phang I, Papadopoulos MC. Intraspinal Pressure Monitoring in a Patient with Spinal Cord Injury Reveals Different Intradural Compartments: Injured Spinal Cord Pressure Evaluation (ISCoPE) Study. Neurocrit Care. 2015 Dec;23(3):414-8. doi: 10.1007/s12028-015-0153-6. PMID 26136148
- [Result] Phang I, Werndle MC, Saadoun S, Varsos G, Czosnyka M, Zoumprouli A, Papadopoulos MC. Expansion duroplasty improves intraspinal pressure, spinal cord perfusion pressure, and vascular pressure reactivity index in patients with traumatic spinal cord injury: injured spinal cord pressure evaluation study. J Neurotrauma. 2015 Jun 15;32(12):865-74. doi: 10.1089/neu.2014.3668. Epub 2015 May 4. PMID 25705999
- [Result] Werndle MC, Saadoun S, Phang I, Czosnyka M, Varsos GV, Czosnyka ZH, Smielewski P, Jamous A, Bell BA, Zoumprouli A, Papadopoulos MC. Monitoring of spinal cord perfusion pressure in acute spinal cord injury: initial findings of the injured spinal cord pressure evaluation study*. Crit Care Med. 2014 Mar;42(3):646-55. doi: 10.1097/CCM.0000000000000028. PMID 24231762
- [Result] Gallagher MJ, Zoumprouli A, Phang I, Schwab JM, Kopp MA, Liebscher T, Papadopoulos MC, Saadoun S. Markedly Deranged Injury Site Metabolism and Impaired Functional Recovery in Acute Spinal Cord Injury Patients With Fever. Crit Care Med. 2018 Jul;46(7):1150-1157. doi: 10.1097/CCM.0000000000003134. PMID 29629987
- [Result] Chen S, Smielewski P, Czosnyka M, Papadopoulos MC, Saadoun S. Continuous Monitoring and Visualization of Optimum Spinal Cord Perfusion Pressure in Patients with Acute Cord Injury. J Neurotrauma. 2017 Nov 1;34(21):2941-2949. doi: 10.1089/neu.2017.4982. Epub 2017 May 24. PMID 28351230
- [Result] Saadoun S, Chen S, Papadopoulos MC. Intraspinal pressure and spinal cord perfusion pressure predict neurological outcome after traumatic spinal cord injury. J Neurol Neurosurg Psychiatry. 2017 May;88(5):452-453. doi: 10.1136/jnnp-2016-314600. Epub 2016 Nov 18. No abstract available. PMID 27864426
- [Result] Chen S, Phang I, Zoumprouli A, Papadopoulos MC, Saadoun S. Metabolic profile of injured human spinal cord determined using surface microdialysis. J Neurochem. 2016 Dec;139(5):700-705. doi: 10.1111/jnc.13854. Epub 2016 Oct 11. PMID 27664973
- [Result] Hogg FRA, Kearney S, Zoumprouli A, Papadopoulos MC, Saadoun S. Acute Spinal Cord Injury: Correlations and Causal Relations Between Intraspinal Pressure, Spinal Cord Perfusion Pressure, Lactate-to-Pyruvate Ratio, and Limb Power. Neurocrit Care. 2021 Feb;34(1):121-129. doi: 10.1007/s12028-020-00988-2. PMID 32435965
- [Result] Gallagher MJ, Hogg FRA, Kearney S, Kopp MA, Blex C, Serdani L, Sherwood O, Schwab JM, Zoumprouli A, Papadopoulos MC, Saadoun S. Effects of local hypothermia-rewarming on physiology, metabolism and inflammation of acutely injured human spinal cord. Sci Rep. 2020 May 15;10(1):8125. doi: 10.1038/s41598-020-64944-y. PMID 32415143
- [Result] Hogg FRA, Gallagher MJ, Kearney S, Zoumprouli A, Papadopoulos MC, Saadoun S. Acute Spinal Cord Injury: Monitoring Lumbar Cerebrospinal Fluid Provides Limited Information about the Injury Site. J Neurotrauma. 2020 May 1;37(9):1156-1164. doi: 10.1089/neu.2019.6789. Epub 2020 Apr 1. PMID 32024422
- [Result] Saadoun S, Papadopoulos MC. Targeted Perfusion Therapy in Spinal Cord Trauma. Neurotherapeutics. 2020 Apr;17(2):511-521. doi: 10.1007/s13311-019-00820-6. PMID 31916236
- [Result] Gallagher MJ, Lopez DM, Sheen HV, Hogg FRA, Zoumprouli A, Papadopoulos MC, Saadoun S. Heterogeneous effect of increasing spinal cord perfusion pressure on sensory evoked potentials recorded from acutely injured human spinal cord. J Crit Care. 2020 Apr;56:145-151. doi: 10.1016/j.jcrc.2019.12.019. Epub 2019 Dec 23. PMID 31901650
- [Result] Gallagher MJ, Hogg FRA, Zoumprouli A, Papadopoulos MC, Saadoun S. Spinal Cord Blood Flow in Patients with Acute Spinal Cord Injuries. J Neurotrauma. 2019 Mar 19;36(6):919-929. doi: 10.1089/neu.2018.5961. Epub 2018 Nov 16. PMID 30351245
- [Result] Hogg FRA, Gallagher MJ, Chen S, Zoumprouli A, Papadopoulos MC, Saadoun S. Predictors of Intraspinal Pressure and Optimal Cord Perfusion Pressure After Traumatic Spinal Cord Injury. Neurocrit Care. 2019 Apr;30(2):421-428. doi: 10.1007/s12028-018-0616-7. PMID 30328047
- [Result] Chen S, Gallagher MJ, Hogg F, Papadopoulos MC, Saadoun S. Visibility Graph Analysis of Intraspinal Pressure Signal Predicts Functional Outcome in Spinal Cord Injured Patients. J Neurotrauma. 2018 Dec 15;35(24):2947-2956. doi: 10.1089/neu.2018.5775. Epub 2018 Sep 27. PMID 30101641
- [Result] Chen S, Gallagher MJ, Papadopoulos MC, Saadoun S. Non-linear Dynamical Analysis of Intraspinal Pressure Signal Predicts Outcome After Spinal Cord Injury. Front Neurol. 2018 Jun 26;9:493. doi: 10.3389/fneur.2018.00493. eCollection 2018. PMID 29997566
- [Derived] Visagan R, Hogg FRA, Gallagher MJ, Kearney S, Zoumprouli A, Papadopoulos MC, Saadoun S. Monitoring Spinal Cord Tissue Oxygen in Patients With Acute, Severe Traumatic Spinal Cord Injuries. Crit Care Med. 2022 May 1;50(5):e477-e486. doi: 10.1097/CCM.0000000000005433. Epub 2022 Jan 6. PMID 35029868